CLINICAL TRIAL: NCT02439593
Title: A Phase II Randomized Study of Concurrent Hyperthermia and Chemoradiotherapy vs. Chemoradiotherapy Alone Following Neoadjuvant Chemotherapy in Locally Advanced Pancreatic Cancer (HEATPAC)
Brief Title: Concurrent Hyperthermia and Chemoradiotherapy in LAPC: Phase II Study
Acronym: HEATPAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Niloy Ranjan Datta, Senior Consultant and Head, Radiation Research, Radiation Oncology, Kantonsspital Aarau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEATPAC
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cancer Pancreas
Keywords: Pancreas; chemoradiotherapy; hyperthermia
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperthermia | interventions — Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: Hyperthermia with chemoradiotherapy vs. Chemoradiotherapy alone
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiotherapy (CTRT) (Control Group) (Active Comparator): Intervention type:
  Drug and Radiation
  Intervention name:
  Drug (Gemcitabine) Radiation (Loco-regional radiotherapy by SIB-IMRT)
  Intervention description:
  Radiotherapy: 5 days a week (Days 1 to 5) of each week for 5.5 weeks (28 fractions), Total dose: 50.4 Gy at 1.8 Gy /fr. over 5.5 weeks Chemotherapy: Gemcitabine (400 mg / sq. m) would be administered weekly 24 hours after hyperthermia on Day 2 and after radiotherapy every week on D2
  Interventions: Other: Chemoradiotherapy (CTRT)
- Thermochemoradiotherapy (CTRTHT) (Experimental): Intervention type:
  Drug, Radiation and Hyperthermia
  Intervention name:
  Drug (Gemcitabine) Radiation (Loco-regional radiotherapy by SIB-IMRT) Hyperthermia (Loco-regional hyperthermia),
  Intervention description:
  Radiotherapy: 5 days a week (Days 1 to 5) of each week for 5.5 weeks (28 fractions), Total dose: 50.4 Gy at 1.8 Gy /fr. over 5.5 weeks Chemotherapy: Gemcitabine (400 mg / sq. m) would be administered weekly 24 hours after hyperthermia on Day 2 and after radiotherapy every week on D2 Hyperthermia: Weekly Local hyperthermia before radiotherapy on D1 of every week, 41-43°C for 60 mins, once every week
  Interventions: Other: Thermochemoradiotherapy (CTRTHT)

INTERVENTIONS:
Other: Chemoradiotherapy (CTRT) — CTRT arm: Locoregional radiotherapy along with concurrent weekly gemcitabine
  Arms: Chemoradiotherapy (CTRT) (Control Group)
Other: Thermochemoradiotherapy (CTRTHT) — Locoregional hyperthermia with concurrent chemoradiotherapy with weekly gemcitabine
  Arms: Thermochemoradiotherapy (CTRTHT)

SUMMARY:
This is a phase II randomized study of concurrent chemoradiotherapy and local hyperthermia (study group) versus chemoradiotherapy alone (control group) following neoadjuvant chemotherapy in locally advanced pancreatic cancer. Each of the treatment arm would have 39 patients based on the expected overall 1 year survival advantage of +20% over the control group (p0=40%).

DETAILED DESCRIPTION:
This phase II randomized trial is a part of the comprehensive protocol designed for the locally advanced pancreatic cancers (LAPC). All patients of LAPC, fulfilling the following criteria of "Unresectable LAPC" would be considered to be eligible for enrolment in the study.

These include:

1. Major venous infiltration / thrombosis of the portal vein or superior mesenteric vein extending for several centimeters (precluding vein resection and reconstruction)
2. Tumor encasement (≥180°) of the superior mesentric artery or proximal hepatic artery
3. Tumor abutment (<180°) of the celiac trunk
4. Tumor invasion of the aorta
5. Presence of metastasis to lymph nodes beyond the field of resection All patients would be reviewed at the Pancreas Cancer Tumor Board, University Hospital Zurich and those fulfilling the above condition/s would be considered for the study protocol of LAPC. Following a detailed work up, all eligible patients with primary tumours more than 4 cm would be considered for HEATPAC study.

Patients would be randomized by random digit using a double blinded strategy into either (a) Control group : Treated with concurrent chemoradiotherapy or (b) Study group: Treated with local hyperthermia along with concurrent chemoradiotherapy.

Treatment in both groups would be initiated with 4 cycles of neo-adjuvant chemotherapy (FOLFIRINOX). At completion of 4 cycles of neo-adjuvant FOLFIRINIOX, patients would be evaluated by PET-CT, 3-4 week following the last cycle of FOLFIRINIOX. Patients in control group would be taken up for concurrent gemcitabine (400 mg / sq.m weekly) along with loco-regional radiotherapy by SIB-IMRT to a dose of 50.4 Gy in 28 fractions. Patients in the study group would be receiving loco-regional hyperthermia to a temperature of 40-41°C, weekly for 1 hour before gemcitabine and before radiotherapy. The gemcitabine and in loco-regional radiotherapy in study group would be similar to that of the control group.

Following the completion of this treatment, patients of both groups would be considered for 8 cycles of adjuvant FOLFIRINOX and followed up with both clinical, heamatological and imaging studies as detailed in the study protocol.

Primary endpoint:

1. Overall survival at 1 year
2. To assess the acute and the late morbidities associated with hyperthermia and chemoradiotherapy in concurrent chemoradiotherapy compared to concurrent chemoradiotherapy alone.

Secondary endpoints:

1. To compare the disease free survival in patients of locally advanced pancreatic cancers following neoadjuvant chemotherapy with FOLOFIRINOX treated with hyperthermia and chemoradiotherapy versus chemoradiotherapy alone.
2. To assess the patterns of failure (both local and systemic) in patients of both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of locally advanced pancreatic cancer with

   * Major venous infiltration / thrombosis of the portal vein or superior mesenteric vein extending for several centimeters
   * Tumor encasement (≥180°) of the superior mesentric artery or proximal hepatic artery
   * Tumor abutment (<180°) of the celiac trunk
   * Tumor invasion of the aorta
   * Presence of metastasis to lymph nodes beyond the field of resection
2. Histopathologically proven ductal adenocarcinoma of the pancreas (biopsy /cytology)
3. Eastern Cooperative Oncology Group (ECOG) performance scale 0 and 1
4. Age: 18 to 80 years
5. At least one of the diameters of the primary tumor or regional lymph node or both should be greater than 4 cm, as confirmed on contrast-enhanced computed tomography (CECT).
6. Patients, have primary tumor or regional lymph node or both lesser than 4 cm, as confirmed on CECT but have specific medical contraindications to stereotactic body radiation therapy or irreversible electroporation or as per patient's preference could be considered for HEATPAC.
7. No evidence of any distant metastasis
8. Patients with microscopic peritoneal carcinomatosis, detected on laparoscopy following 4 cycles on neo-adjuvant FOLFIRINOX would be included.
9. Estimated life expectancy of at least 6 months
10. Adequate kidney functionality defined as creatinine clearance >50ml/min
11. Adequate liver functionality defined as total bilirubin ≤ 2x of the upper limit of normal
12. Adequate bone marrow reserves: White blood cell count ≥ 2.5 x 10˄9/L, Platelet count ≥ 100 x 10˄9/L, Hemoglobin ≥ 8.0g/L
13. Women of child-bearing age must secure sufficient contraception control during the clinical trial and six months after the clinical trial is completed
14. For females of child bearing potential, negative pregnancy test within 2 week prior to randomization.
15. Female patients should not be lactating
16. Absence of psychological, familial, sociological or geographical condition that could potentially hamper compliance with the study protocol and follow-up schedule

Exclusion Criteria:

1. Histopathology other than ductal adenocarcinoma pancreas
2. Prior radiotherapy to the site of treatment
3. Patients with unequivocal distant metastasis including liver
4. Patients with gross peritoneal carcinomatosis on laparoscopy
5. No prior or concurrent malignancies other than surgically treated squamous cell or basal cell carcinoma of the skin
6. No serious medical illness which would prevent informed consent or limit survival to less than 2 years
7. Active uncontrolled bacterial, viral or fungal infections until these conditions are corrected or controlled.
8. Psychiatric or addictive disorders or other conditions that would preclude the patient from meeting the study requirements.
9. Patients having metal implants, pacemakers or clustered markers.
10. Metallic endobiliary stenting would be a contraindication, hence plastic stents may be used if biliary drainage is indicated.
11. Patient with a history of myocardial infarction within the past 12 months
12. No connective disease disorders that contraindicate radiotherapy, e.g., Scleroderma
13. Pre-existing grade 2 peripheral neuropathy
14. Any known contraindication or hypersensitivity to the chemotherapeutic agents
15. Pregnancy, lactation period or lack of reliable contraception
16. Any other disease or therapy, which, present a risk to the patient or which are not compatible with the aims of the clinical trial
17. Patients would express their inability to travel on their own to Kantonsspital Aarau, (KSA) for hyperthermia treatment
18. Indications that the person concerned will be noncompliant to the clinical trial plan because of unwillingness to cooperate or difficulties in keeping the check-up appointments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (at 1 year) | From date of randomization until the date of death from any cause assesed at 1 year or whichever is earlier
  Overall survival

SECONDARY OUTCOMES:
Progression free survival (as per Response Evaluation Criteria in Solid Tumours (RECIST), v1.1) | From date of randomization until the first docemented disease progression as evident on CECT / PET-CT / MRI as per RECIST criteria (v1.1), whichever came first assessed upto the end of study period of 60 weeks
  Progression free survival
Patterns of failure : both local and systemic (as per RECIST, v1.1) | From date of randomization until the disease progression either locally or at distant sites as evident on CECT / PET-CT / MRI as per RECIST criteria (v1.1), whichever came first assessed upto the end of study period of 60 weeks
  Patterns of failure : both local and systemic
Acute and late morbidity (as per Common Toxicity Criteria for Adverse Effects (CTCAE) v4.03) | Acute or late morbidity from date of randomization until the patients death from any cause as per the CTCAE v4.03 whichever came first assessed upto the end of study period of 60 weeks
  Acute and late morbidity that are ascribed to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Niloy R Datta, MD,DNB, Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Derived] Datta NR, Pestalozzi B, Clavien PA, Siebenhuner A, Puric E, Khan S, Mamot C, Riesterer O, Knuchel J, Reiner CS, Bodis S; members of the HEATPAC Trial Group. "HEATPAC" - a phase II randomized study of concurrent thermochemoradiotherapy versus chemoradiotherapy alone in locally advanced pancreatic cancer. Radiat Oncol. 2017 Nov 21;12(1):183. doi: 10.1186/s13014-017-0923-8. PMID 29162142